CLINICAL TRIAL: NCT06802874
Title: Maternal-fetal Outcomes of Genital Blood Loss Beyond 18 Weeks of Pregnancy
Acronym: PEG18
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PEG18
Record Dates: First submitted 2024-12-30; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Blood Loss
Keywords: Pregnancy blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective is to assess in terms of frequency the adverse outcomes (premature birth, maternal-fetal haemorrhage, maternal fetal-neonatal death) of pregnancies of women attending the obstetric-gynaecological emergency department for genital bleeding beyond the 18th week of pregnancy.

DETAILED DESCRIPTION:
The investigators decided to conduct this study because it is important on the one hand to carefully evaluate maternal-fetal outcomes in pregnancies characterised by genital bleeding in the second and third trimesters and on the other hand to evaluate the sonographic diagnostic capacity for identifying the aetiology of these genital bleedings, in order to understand whether the possibility of identifying a specific cause of the bleeding has also improved over time as sonographic techniques have improved. This could then allow management and subsequent obstetrical controls to be adapted in a more accurate and indivudualised manner.

For the purpose of this study, no study-specific visits are planned. Data collected during pregnancy and delivery data for patients who gave birth at our centre will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy beyond 18 weeks gestational age complicated by genital bleeding;
* Age of the patient ≥18 years;
* Delivery at the O.U. of Obstetrics and Prenatal Age Medicine

Exclusion Criteria:

None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include pregnant patients over 18 weeks of pregnancy referred to the obstetrical emergency department of the division of Obstetrics and Prenatal Age Medicine of IRCCS Azienda Ospedaliero Universitaria di Bologna for genital blood loss.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of hospitalization for genital blood loss | After the 18th week of pregnancy
Percentage of preterm births | After delivery, up to 24 weeks
Percentage of spontaneous deliveries, operative vaginal, cesarean sections (elective, urgent, emergent) | After delivery, up to 24 weeks
Frequency of antihemorrhagic therapy and maternal transfusions | Intra-partum and post-partum, up to 24 weeks
Frequency of live births, average APGAR, average pH of umbilical artery or vein, average neonatal weight | After delivery, up to 24 weeks
Average length of hospitalization in hours | During Hospitalization, up to 24 weeks

SECONDARY OUTCOMES:
Frequency of finding abnormal ultrasound findings corresponding to the etiology of bleeding | During the obstetric ultrasound performed at the time of admission
  To assess whether the ultrasound capability in detecting a specific etiology of bleeding has improved over time in conjunction with the evolution of technology and resolution of ultrasound equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Morganti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy